CLINICAL TRIAL: NCT05096728
Title: Frequency and Dosing of Long Acting Anti-Hypertensive Agent in Women With Pre-eclampsia With Severe Features Undergoing Expectant Management: A Randomized Controlled Trial
Brief Title: Nifedipine Dosing Daily vs Twice a Day for Pre-eclampsia With Severe Features (NOPPI)
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Kara M Rood, MD, Assistant Professor, Ohio State University
Other Study IDs: 2021H0292
Record Dates: First submitted 2021-09-17; First posted 2021-10-27 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Preeclampsia With Severe Features
Keywords: preeclampsia severe; Nifedipine XL 60mg; Nifedipine XL 30mg
MeSH Terms: interventions — Nifedipine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Once daily Nifedipine XL 60mg: Participants will receive Nifedipine XL once daily 60 mg for 48 hours.
  Interventions: Drug: Nifedipine XL
- Twice daily Nifedipine XL 30mg: Participants will receive Nifedipine XL twice daily 30 mg for 48 hours.
  Interventions: Drug: Nifedipine XL

INTERVENTIONS:
Drug: Nifedipine XL — Patients will be enrolled when the primary provider has made the decision to increase the patient's daily dose of Procardia XL from 30mg to 60mg. Participants will be randomized in to one of two groups
  * Once daily Nifedipine XL 60mg Vs.
  * Twice daily Nifedipine XL 30mg
  Other Names: Procardia XL

SUMMARY:
The investigators propose a randomized controlled unblinded trial to evaluate rates of optimal blood pressure control between Nifedipine 60mg XL once daily vs. Nifedipine 30mg XL twice daily in patients admitted for expectant management with pre-eclampsia with severe features. Patients will be approached for consent when they are placed on 30mg of Nifedipine daily by their primary provider and will be enrolled in the study when the primary provider has made the decision to increase the patient's daily dose of Nifedipine XL from 30mg to 60mg.

DETAILED DESCRIPTION:
This is a randomized controlled unblinded trial at The Ohio State University comparing Nifedipine XL 60mg daily to 30mg twice daily in patients admitted for expectant management for pre-eclampsia with severe features.

Potential study participants will be identified at the time of admission to the antepartum unit. Inclusion criteria must be met, namely patient's age, gestational age, diagnosis of preeclampsia with severe features.

Patients will be approached for consent when they are placed on 30mg of Nifedipine daily by their primary provider and will be enrolled in the study when the primary provider has made the decision to increase the patient's daily dose of Nifedipine XL from 30mg to 60mg. Participants will be randomized in to one of two groups:

* Once daily Nifedipine XL 60mg Vs.
* Twice daily Nifedipine XL 30mg

Once enrolled and randomized, blood pressures will be monitored every 4 hours as is standard on the antepartum unit. Blood pressures for the primary outcome will be collected 24 hours after the patient is randomized and initiated on their above regimen. This is to allow the medication to reach steady state prior to collected information on optimal blood pressures. The primary outcome will consist of blood pressure values collected q4 hours beginning 24h-48h after receiving their first dose of the randomized dose regimen.

Algorithms for the administration of intravenous labetalol, Nifedipine or hydralazine will be utilized by the primary provider at his or her discretion.

Women may take the medication concurrently with intravenous labetalol, hydralazine, or immediate release Nifedipine for the treatment of severe blood pressures as determined by their primary provider.

All other obstetric care will be at the discretion of the primary provider, including but not limited to addition of second long-acting hypertensive agents, decision to proceed with delivery, IV magnesium for seizure prophylaxis and recommendations regarding mode of delivery. Data will be collected on these components of routine obstetric care. Analysis will be by intent to treat.

A subset of patients will be enrolled for a pharmacokinetic study and blood will be collected at prespecified times following administration of the randomized Nifedipine XL regimen.

ELIGIBILITY:
Inclusion Criteria:

* Women age 18-45 with a viable single or twin intrauterine pregnancy between 22 0/7 and 33 6/7 weeks gestation based on the best obstetric estimate by ACOG criteria.
* Undergoing expectant management for a diagnosis of preeclampsia with severe features and already initiated on 30mg Nifedipine XL. The patient may or may not have already received acute treatment for severe blood pressures.

Exclusion Criteria:

* Known allergy or adverse reaction to Nifedipine or any medical condition where Nifedipine is contraindicated, such as galactose intolerance, severe GI stricture, and GI hypomotility disorder.
* Participation in another trial without prior approval
* Currently receiving a daily dose of Nifedipine XL of 60mg or greater
* Continuation of alternate long-acting anti-hypertensive medication on admission
* Physician/provider or patient refusal
* Triplet or higher order pregnancy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Pregnant women undergoing expectant management for a diagnosis of preeclampsia with severe features already initiated on 30mg Nifedipine XL and the primary provider has made the decision to increase the patient's daily dose of Procardia XL from 30mg to 60mg. .
Sampling Method: Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-12-06 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Comparing the rates of suboptimal blood pressure | on day 2 (24 hour-48 hour) after the patient has been enrolled
  Comparing the rates of suboptimal blood pressure, defined as frequency of systolic >150 mmHg and/or diastolic >100 mmHg blood pressure. Blood pressure measurements will be measured every 4 hours on day 2 (24 hour-48 hour) after the patient has been enrolled, randomized, and initiated on either once daily Nifedipine XL 60mg or twice daily Nifedipine XL 30mg.

SECONDARY OUTCOMES:
Evaluating mean systolic and diastolic blood pressure and mean arterial pressure | on day 2 (24 hour-48 hour) after the patient has been enrolled
  Evaluating mean systolic and diastolic blood pressure and mean arterial pressure measured on day 2 (24h-48h) after the patient has been enrolled, randomized, and initiated on Nifedipine regimen
Evaluating concentration of Nifedipine in blood | on day 2 (24 hour-48 hour) after the patient has been enrolled
  Evaluating concentration of Nifedipine in blood measured at prespecified times taken on day 2 (24 hour-48 hour) after the patient has been enrolled, randomized, and initiated on a Nifedipine regimen
Evaluating number of route of delivery | Through study completion, an average of 2 years
Evaluating number of days in expectant management from enrollment | Through study completion, an average of 2 years
Evaluating frequency of indications for cesarean section | Through study completion, an average of 2 years
Evaluating frequency of need for acute acting anti-hypertensive treatment (IR Nifedipine, IV labetalol, or IV hydralazine) | on day 2 (24 hour-48 hour) after the patient has been enrolled
Evaluating number of delivery less than 34 weeks | Through study completion, an average of 2 years
Evaluating gestational age at delivery | Through study completion, an average of 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Kara Rood, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center OB/GYN Maternal and Fetal Medicine, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No